CLINICAL TRIAL: NCT01474213
Title: Dexmedetomidine Versus Remifentanil Target Controlled Infusion for Sedation During Awake Fibreoptic Nasotracheal Intubation
Brief Title: Sedation Effect of Dexmedetomidine Versus Remifentanil to Fibreoptic Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Rong Hu, consultant in anesthesilogy department of Shanghai 9th People's Hospital, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: JYMZK-002
Record Dates: First submitted 2011-10-31; First posted 2011-11-18 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: Intubation; Difficult
Keywords: dexmedetomidine; remifentanil; awake nasotracheal fibreoptic intubation; oral maxillofacial surgery; difficult airway; adult
MeSH Terms: interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmedetomidine (Active Comparator): a loading dose (1.5mcg/kg) infused over10 min followed by a continuous infusion of 0.7 μg/kg/h
  Interventions: Drug: dexmedetomidine group
- remifentanil (Active Comparator): The initial target was 3.0 ng/ml and the TCI was adjusted by 0.5 ng/ml after the target concentration at the effect site had equilibrated with the plasma concentration, until the desired level of sedation was acheived.
  Interventions: Drug: remifentanil group

INTERVENTIONS:
Drug: dexmedetomidine group — 1-1.5cmg/kg dexmedetomidine infusion within 10 minutes, while followed by maintainly infusing 0.7cmg/kg/min dexmedetomidine
  Other Names: Dexmedetomidine Hydrochloride Injection
  Arms: dexmedetomidine
Drug: remifentanil group — target controlled 3.5-4ng/ml remifentanil infused(blood plasma concentration)
  Other Names: Remifentanil
  Arms: remifentanil

SUMMARY:
The purpose of this study is to compare the sedation effect of dexmedetomidine and target controlled remifentanil for awake nasotracheal fibreoptic intubation in patients undergoing oral maxillofacial surgery.

DETAILED DESCRIPTION:
Awake fibreoptic nasotracheal intubation is an effective technique for the management of patients with difficult airways undergoing oral maxillofacial surgery. Both optimal intubating conditions and patient comfort are paramount while preparing the patient for fibreoptic intubation. One challenge associated with procedure is to provide adequate sedation while maintaining patients' airway ventilation. Dexmedetomidine, because of its sedative,analgesic properties and minimal influence on patients' ventilation, might be a useful management for it. While with the development of target controlled infusion (TCI) technology, remifentanil sedation becomes a potential sedation in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-III adult patients with difficult airway, who were undergoing elective oral maxillofacial surgery

Exclusion Criteria:

* pregnant or lactating female,
* long-term opioids or sedative medication,
* patients < 18 years of age,
* severe bradycardia (HR < 50 beats/min),
* hypotension (systolic pressure < 90mmHg),
* any type of atrioventricular block on the ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, MD, PHD, Study Chair — Anesthesiology Department, Shanghai Ninth People's Hospital Affiliated Shanghai JiaoTong University School of Medicine
Locations (2):
- China (2):
  - Shanghai JiaoTong University, School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty two adult patients, American Society of Anesthesiologist (ASA) score of I-III, were recruited for an elective awake fibreoptic nasotracheal intubation due to the diagnosis of maxillofacial cancer or fracture with limited mouth opening
Pre-assignment Details: One patient declined consent and one operation was cancelled.
Groups:
- Dexmedetomidine Infusion for Sedation: Patients in the dexmedetomidine group received a loading dose (1.5 μg kg-1) infused over10 min followed by a continuous infusion of 0.7 μg kg-1 h-1.
- Remifentanil Target Controlled Infusion: Patients in the remifentanil group received remifentanil via an Orchestra Base Primea (Fresenius Vial) infusion system using a Minto pharmacokinetic model. The initial target was 3.0 ng ml-1 and the TCI was adjusted by 0.5 ng ml-1 after the target concentration at the effect site had equilibrated with the plasma concentration, until the desired level of sedation was reached.
Period: Overall Study
Arm/Group | Dexmedetomidine Infusion for Sedation | Remifentanil Target Controlled Infusion
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Infusion for Sedation | Remifentanil Target Controlled Infusion | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.4 (15.2) | 37.8 (14.9) | 38.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  China | 20 | 20 | 40

OUTCOME MEASURES:

1. Secondary Outcome: Patient's Reaction to Procedure
Description: Ramsay score during the endoscopy intubation from 1 to 6. The higher scores means the deeper sedation level.
  Clinical score Level of sedation
  1. Patient is anxious and agitated or restless, or both
  2. Patient is cooperative, oriented and tranquil
  3. Patient responds to commands only
  4. Patient exhibits a brisk response to a light glabellar (between the eyebrows) tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to a light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response to stimuli
Time Frame: the duration of intubation, an expected average of 10 minutes
Population: Power calculation identified a minimum requirement of 15 patients randomized to each group to demonstrate a 20% difference in outcome scores with a power of 0.8 and a type I error of 0.05 according to our preliminary study.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Remifetanil Target Controlled Infusion: Patients in the remifentanil group received remifentanil via an Orchestra Base Primea (Fresenius Vial) infusion system using a Minto pharmacokinetic model. The initial target was 3.0 ng ml-1 and the TCI was adjusted by 0.5 ng ml-1 after the target concentration at the effect site had equilibrated with the plasma concentration, until the desired level of sedation was reached.
- Dexmedetomidine Continuously Infusion for Sedation: Patients in the dexmedetomidine group received a loading dose (1.5 μg kg-1) infused over10 min followed by a continuous infusion of 0.7 μg kg-1 h-1.
Arm/Group | Remifetanil Target Controlled Infusion | Dexmedetomidine Continuously Infusion for Sedation
Number analyzed (Participants) | 20 | 20
units on a scale | 3 [2 to 4] | 3 [2 to 4]

2. Secondary Outcome: Post Operative Visit
Description: visit the patients to ensure their memory of intubation. Postoperative interview asked the patients' memory of the fiberoptic intubation Amnesia Recall of endoscopy Yes No Recall of intubation Yes No The number is the patients who remember the operation procedure.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Remifetanil Target Controlled Infusion | Dexmedetomidine Continuously Infusion for Sedation
Number analyzed (Participants) | 20 | 20
participants | 13 | 6

3. Secondary Outcome: Mean Arterial Blood Pressure
Description: MAP at 15 minutes before intuation, endoscopy point and intubation point between two groups were compared.
Time Frame: 15 minutes before intubation, endoscopy point, intubation point
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Remifetanil Target Controlled Infusion | Dexmedetomidine Continuously Infusion for Sedation
Number analyzed (Participants) | 20 | 20
mmHg
  MAP at intubation point | 101.3 (14.5) | 103.5 (9.9)
  MAP at 15 minutes before intubation | 93.8 (10.0) | 90.4 (10.6)
  MAP at endoscopy point | 102.8 (10.5) | 99.5 (10.7)

4. Secondary Outcome: Heart Rate
Description: Heart rate at 15 minutes before intuation, endoscopy point and intubation point between two groups were compared.
Time Frame: 15 minutes before intubation, endoscopy point, intubation point
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Remifetanil Target Controlled Infusion | Dexmedetomidine Continuously Infusion for Sedation
Number analyzed (Participants) | 20 | 20
beats per minute
  Heart rate15 minutes before intubation | 76.4 (11.7) | 72.8 (10.2)
  Heart rate at endoscopy point | 76.9 (15.9) | 56.5 (9.5)
  Heart rate at intubation point | 77.8 (15.3) | 65.4 (9.8)

5. Secondary Outcome: Peripheral Oxygen Saturation(SPO2)
Description: Peripheral oxygen saturation at 15 minutes before intuation, endoscopy point and intubation point between two groups were compared.
Time Frame: 15 minutes before intubation, endoscopy point, intubation point
Measure: Mean (Standard Deviation); unit: percentage oxygen saturation
Arm/Group | Remifetanil Target Controlled Infusion | Dexmedetomidine Continuously Infusion for Sedation
Number analyzed (Participants) | 20 | 20
percentage oxygen saturation
  15 minutes before intubation | 99.0 (1.2) [8 to 19] | 98.9 (1.1) [9 to 17]
  at endoscopy point | 95.8 (2.6) | 98.2 (2.0)
  at intubation point | 98.2 (1.9) | 99.0 (1.4)

6. Secondary Outcome: Cardiac Rhythm
Description: Number of Participants with Abnormal Cardiac Rhythm(including any type of the abnormal cardiac rhythm from 15 minutes before intubation and during the intubation procedure was recorded such as sinus arrhythm, atrial or ventricular premature beats and atrioventricular block) was recorded.
Time Frame: 15 minutes before intubation and duration of intubation
Measure: Number; unit: participants
Groups:
- Remifetanil Target Controlled Infusion: Two patients in remifentanil group exhibited bradycardia(heart rate<50beats per minute) during endoscopy and intubation period.
- Dexmedetomidine Continuously Infusion for Sedation: Three patients in dexmedetomidine group exhibited bradycardia(heart rate<50beats per minute) during endoscopy and intubation period.
Arm/Group | Remifetanil Target Controlled Infusion | Dexmedetomidine Continuously Infusion for Sedation
Number analyzed (Participants) | 20 | 20
participants | 2 | 3

7. Primary Outcome: Endoscopy Scores
Description: Endoscopy was graded from 0 to 5, with lower scores indicating a possibly better condition.
  Endoscopy score 0 1 2 3 4 5: 1)Grimacing 2)localising 3)Coughing on lignocaine via scope 4)Coughing on entering infraglottic space 5)Prolonged coughing
Time Frame: during the procedure of fibreoptic and tracheal intubation
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Remifentanil Target Controlled Infusion: Patients in the remifentanil group received remifentanil via an Orchestra Base Primea (Fresenius Vial) infusion system using a Minto pharmacokinetic model. The initial target was 3.0 ng ml-1 and the TCI was adjusted by 0.5 ng ml-1 after the target concentration at the effect site (had equilibrated with the plasma concentration, until the desired level of sedation was reached.
Arm/Group | Remifentanil Target Controlled Infusion | Dexmedetomidine Infusion for Sedation
Number analyzed (Participants) | 20 | 20
units on a scale | 3 [1 to 3] | 2 [0 to 3]

8. Primary Outcome: Intubation Score
Description: graded from 0 to 5, with lower scores indicating better conditions Intubation score 0 1 2 3 4 5: 1)Grimacing when tube in nares 2)Localising with one limb at any stage 3)Localising with two limbs at any stage 4)Coughing on entering trachea 5)Prolonged coughing
Time Frame: during the inserting of the tracheal tube
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remifetanil Target Controlled Infusion | Dexmedetomidine Continuously Infusion for Sedation
Number analyzed (Participants) | 20 | 20
units on a scale | 1 [1 to 3] | 1 [0 to 3]

9. Secondary Outcome: Post Intubation Score
Description: Post-intubation was scored from 1 to 3, with higher scores indicating a worse outcome.
  Post-intubation score 1 2 3
  1. Cooperative, obeying commands
  2. Uncomfortable, GA imminent
  3. Other（specify）
Time Frame: immediately after the intubation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remifetanil Target Controlled Infusion | Dexmedetomidine Continuously Infusion for Sedation
Number analyzed (Participants) | 20 | 20
units on a scale | 1 [1 to 3] | 1 [1 to 2]

ADVERSE EVENTS:
Time Frame: during the endoscopy and intubation period
Arm/Group | Dexmedetomidine Infusion for Sedation | Remifentanil Target Controlled Infusion
Serious Adverse Events (participants affected / at risk) | 3/20 | 2/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine Infusion for Sedation (N=20) | Remifentanil Target Controlled Infusion (N=20)
bradycardia (Cardiac disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
The sample number is relatively small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes